CLINICAL TRIAL: NCT04972253
Title: Biomarker-directed Neoadjuvant Therapy for Cisplatin-ineligible or Cisplatin-refusing Muscle-invasive Bladder Cancer: Phase I Bladder Cancer Signal Seeking Trial
Brief Title: Phase I BLASST-3 Trial
Acronym: (BLASST)-3
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Guru P. Sonpavde (Other)
Collaborators: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor-Investigator, Guru P. Sonpavde, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-162
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Bladder Transitional Cell Carcinoma; Bladder Cancer; Fibroblast Growth Factor Receptor
Keywords: Bladder transitional cell carcinoma; Bladder Cancer; Fibroblast growth factor receptor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Acrocephalosyndactylia | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infigratinib (Experimental): * Infigratinib daily dosage per protocol 3-week on/1-week off schedule. 4 weeks will constitute 1 cycle of therapy.
  * Participants will receive 2 cycles (i.e. 8 weeks) and the treatment will be administered as an outpatient.
  * After completion of therapy, patients will undergo a CT of the chest, abdomen and pelvis (within 2 weeks of the last dose of therapy) and then proceed to Radical cystectomy 2-4 weeks after the last dose of therapy.
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Oral, dosage per protocol
  Other Names: BGJ-398

SUMMARY:
The aim of this research is to see whether using a drug that blocks a protein called FGFR (fibroblast growth factor receptor) prior to surgery is safe and effective in patients with bladder cancer that have mutations in FGFR3 or FGFR2 and who cannot receive chemotherapy with cisplatin prior to surgery

The name of the study drug involved in this study is:

- Infigratinib

DETAILED DESCRIPTION:
This is a single-center (DF/HCC) prospective feasibility study to assess biomarker-directed neoadjuvant therapy in patients with cT2-T4aN0 MIBC who are candidates for radical cystectomy (RC) and ineligible for, or refuse, cisplatin-based neoadjuvant chemotherapy (NAC).

This research study involves using a drug that inhibits FGFR in patients with bladder cancer (that have mutations in FGFR) prior to surgery.

The name of the study drug involved in this study is:

- Infigratinib

The research study procedures include pre-screening for eligibility and study treatment including evaluations and follow up visits. This pre-screening is already done as clinical care. Study participants will receive study treatment for 2 months prior to surgery and will be followed for at least 1 year after undergoing surgery.

It is expected that about 12 people will take part in this research study.

This research study is a Phase I clinical trial, which tests the safety of an investigational drug (infigratinib) and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

This research study is also a Feasibility Study, which is the first time investigators are examining this drug in patients with bladder cancer that has not spread to other organs. The U.S. Food and Drug Administration (FDA) has not approved infigratinib as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g. HIPAA) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
* Age ≥ 18 years at time of study entry (no safety data in pediatric patients is available for infigratinib).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (See Appendix A).
* Histologically confirmed bladder transitional cell carcinoma (TCC)

  -- Patients with mixed histology are required to have a component of TCC, and no component of small cell histology
* cT2-T4a N0 M0 disease after radiographic staging of chest, abdomen and pelvis, considered appropriate and planned for radical cystectomy as assessed by a Urologic Oncologist.
* Presence of the following FGFR3/2 activating alterations, as detected by either plasma or urine cfDNA or cfRNA or by tissue-based NGS (Predicine, Hayward, CA):

  * Mutations in exon 7 (R248C, S249C)
  * Mutations in exon 10 (G372C, A393E, Y375C)
  * Mutations in exon 15 (K652M/T, K652E/Q)
  * Any FGFR3/2 gene fusion (Availability of baseline archival tumor tissue for identification of FGFR3/2 alterations is not required, but tissue will be obtained when available including either FFPE tumor tissue block or a minimum of fifteen 5μm unstained FFPE slides and fifteen 10μm unstained FFPE slides with an associated pathology report is required)
* Ineligibility for cisplatin-based chemotherapy, defined by any of the following:

  * Creatinine clearance (CL) <60 mL/min. GFR should be calculated from serum/plasma creatinine using the Cockcroft-Gault formula.
  * CTCAE v5.0 Grade > 1 hearing loss
  * CTCAE v5.0 Grade > 1 neuropathy
  * NYHA Class > II cardiac dysfunction
  * Patients not meeting the above criteria are eligible if he/she declines neoadjuvant cisplatin-based chemotherapy after specific informed consent describing the known benefits of cisplatin-based chemotherapy. The reason for cisplatin-ineligibility based on the above criteria or cisplatin refusal should be documented on the case report form.
* Adequate organ function laboratory values as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
  * Platelet count ≥100 x 109/L (>75,000 per mm3)
  * International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) < 1.5 x ULN, unless the patient is receiving anticoagulation therapy provided INR or PTT is within the therapeutic range of the intended anticoagulant therapy.
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)

  -- This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT)/ALT (SGPT) ≤1.5 x institutional upper limit of normal
* Measured creatinine CL >30 mL/min or Calculated creatinine CL>30 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance:

  * Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age)/72 x serum creatinine (mg/dL)
  * Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85/ 72 x serum creatinine (mg/dL)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following agespecific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient has ability and willingness to sign a written informed consent document and is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Patients with primary TCC of the ureter, urethra, or renal pelvis without TCC of the bladder
* Inoperable tumor(s) with fixation to the pelvic wall on clinical exam
* Any previous systemic chemotherapy or radiotherapy for TCC of bladder
* Participation in another clinical study with an investigational product during the last 6 months
* Any prior participation in a study involving an FGFR inhibitor.
* Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (e.g. cervical cancer in situ)
* Receipt of the last dose of intravesical chemotherapy or biologic therapy ≤ 42 days (6 weeks) prior to the first dose of study drug for patients who have received prior intravesical chemotherapy or biologic therapy (e.g. BCG)
* Any unresolved toxicity NCI CTCAE version 5.0 Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients currently receiving treatment with drugs that are known to be strong CYP3A4 inducers or inhibitors, including anti-epileptic drugs.
* Use of medications that are known to prolong the QT interval and/or associated with a risk of torsade de pointes 7 days prior to the first dose of infigratinib.
* Use of amiodarone within 90 days prior to first dose of infigratinib.
* Use of medications that increase serum levels of calcium and/or phosphorus.
* Concurrent use of warfarin or other coumadin-derivative anticoagulants; heparin and/or low molecular-weight heparins are permitted.
* Inorganic phosphorus and/or total/ionized serum calcium outside normal limits prior to study entry.
* Have clinically significant cardiac disease, including any of the following:

  * New York Heart Association (NYHA) Class ≥2B; subjects with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the NYHA classification.
  * Presence of Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≥2 ventricular arrhythmias, atrial fibrillation, bradycardia, or conduction abnormality
  * Unstable angina pectoris or acute myocardial infarction ≤3 months prior to first dose of study drug
  * QTcF >470 msec (males and females). Note: If the QTcF is >470 msec in the first ECG, a total of 3 ECGs separated by at least 5 minutes should be performed. If the average of these 3 consecutive results for QTcF is ≤470 msec, the subject meets eligibility in this regard
  * Known history of congenital long QT syndrome.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of infigratinib. NB: local surgery of isolated lesions for palliative intent is acceptable.
* History of allogeneic organ transplantation
* Current evidence of corneal or retinal disorder/keratopathy
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Female patients who are pregnant or breastfeeding, or patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of infigratinib monotherapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Inability to swallow oral medications
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
≥ 70% of patients receiving at least 1 dose of study treatment followed by completion of radical cystectomy (Feasibility) | time of first administration of study treatment until 4 weeks after RC up to 3 months
  Feasibility is defined as ≥ 70% of patients receiving at least 1 dose of study treatment followed by completion of radical cystectomy in the absence of DLT up to 4 weeks post-RC.
  Dose-limiting toxicities (DLTs) will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria). DLT will be defined as an adverse event (AE) or abnormal laboratory value deemed related to therapy with infigratinib, including those AEs and abnormal laboratory values that result in a failure to meet the criteria for re-treatment.

SECONDARY OUTCOMES:
Pathologic response (<ypT2N0) at time of RC. | 3 months
  Pathologic response is defined as <pT2N0 disease at the time of RC (e.g. pT0N0, pT1N0, pTaN0, or pTisN0)
Pathologic complete response (pCR) at time of RC. | 3 months
  Pathologic complete response (pCR) is defined as achievement of pT0N0 disease at RC.
Relapse-free survival (RFS) after RC. | 4 weeks after end of treatment, then every 12-24 weeks up to 1 year
  Relapse-free survival (RFS) is defined as the duration of time from time of RC to time of documented disease relapse or recurrence after RC, or death from any cause. Patients who have received at least one cycle of therapy and have undergone RC will be considered evaluable for RFS.
Progression-free proportion after neoadjuvant infigratinib, prior to RC | 2 months
  Progression prior to RC will be defined as radiologic progression by RECIST 1.1 with development of radiologic T4b and/or N1/N2/N3 and/or or M1 disease (per RECIST 1.1) in scans obtained after commencement of neoadjuvant therapy and prior to RC

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu